CLINICAL TRIAL: NCT05442957
Title: A Multi-Site, Parallel-Group, Randomized Clinical Trial Comparing a Brief Tele-Cognitive Behavioral Therapy Intervention (BRIGHT) With Attention Control for the Reduction of Body Image-Related Distress Among Head and Neck Cancer Survivors
Brief Title: Building a Renewed ImaGe After Head & Neck Cancer Treatment (BRIGHT) Multi-Site RCT
Acronym: BRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Graboyes, Associate Professor, Department of Otolaryngology- Head and Neck Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO 00110248; R37CA269385 (NIH)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Body Image Disturbance; Body Image; Survivorship; Psychosocial Impairment; Mental Health Issue
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIGHT (Experimental): BRIGHT is a manualized theory-based video tele-cognitive behavioral therapy (CBT) intervention delivered one-on-one by a licensed clinical psychologist.
  Interventions: Behavioral: BRIGHT
- Attention Control (Active Comparator): The attention control arm is a manualized video tele-supportive care intervention that addresses non-body image aspects of HNC survivorship.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: BRIGHT — BRIGHT is a manualized theory-based tele-CBT intervention consisting of 6 weekly 60-minute sessions. BRIGHT is delivered one-on-one by a licensed clinical psychologist at each site via standard video tele-CBT platform. BRIGHT session topics include (1) psychoeducation about the cognitive model of body image, (2) self-monitoring about thoughts, feelings, and body image behaviors, (3) cognitive restructuring to identify and challenge unhelpful automatic HNC body image thoughts, (4) positive body image coping strategies, (5) social support and identifying personal value, and (6) thinking ahead and planning for setbacks.
  Arms: BRIGHT
Behavioral: Attention Control — AC is a manualized video-tele-supportive care intervention that addresses non-body image aspects of HNC survivorship. Identical to BRIGHT, AC consists of 6 weekly 60-minute sessions delivered by a trained empathic interventionist via standard video-telemedicine platform. AC session topics include (1) Introduction to HNC survivorship, (2) Post-Treatment Side Effects (3) Psychosocial Aspects of HNC, (4) Health Promotion and Nutritional Challenges, (5) Financial Distress and Return to Work, and (6) Cancer Recurrence. AC controls for professional attention (i.e., ensuring that findings are not driven by simply interacting with an empathic interventionist), common factors, dose, and delivery method while not providing the active, behavior change mechanism in BRIGHT.
  Arms: Attention Control

SUMMARY:
In this multi-center randomized clinical trial, head and neck cancer (HNC) survivors with clinically significant body image distress (BID) (N=180) will be randomized to BRIGHT (a brief video tele-cognitive behavioral therapy intervention) or Attention Control (AC, a manualized tele-supportive care intervention that controls for professional attention, dose, delivery method, and common factors). HNC survivors will complete IMAGE-HN (a validated patient-reported outcome measure [PROM] of HNC-related body image distress [BID]; primary endpoint), measures of psychological and social well-being and quality of life (QOL), and measures of theory-derived mechanisms of change underlying BRIGHT (mediators).

DETAILED DESCRIPTION:
We will perform a multi-site randomized clinical trial (RCT) comparing BRIGHT with AC to test our hypotheses that BRIGHT reduces BID and improves psychological and social well-being and QOL at 2, 3, 6, and 9-months post-randomization by enhancing body image coping skills and decreasing unhelpful automatic thoughts. HNC survivors with clinically significant BID (N=180) from multiple sites in the United States will be randomized 1:1 to BRIGHT or AC. We will conduct semi-structured interviews with key stakeholders (n=10/site) and in-depth site visits to assess barriers and facilitators of the adoption of BRIGHT and develop an implementation toolkit to enhance the future adoption of BRIGHT into routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years on the day of informed consent
2. History of pathologically confirmed squamous cell carcinoma (or histologic variant) of the oral cavity, pharynx, larynx, nose/paranasal sinuses, carcinoma of a major or minor salivary gland, or cutaneous malignancy of the face or neck
3. History of curative intent surgery with or without adjuvant therapy, with or without reconstruction
4. Completion of oncologic treatment within 12 months of study enrollment (but no sooner than 6 weeks post-treatment completion)

   1. Patients who complete definitive HNC-directed therapy (e.g., surgery or radiation therapy) but are on adjuvant immunotherapy are considered eligible
   2. Oncologic treatment refers to cancer-directed therapy; non-cancer surgery (e.g., trachea-esophageal puncture, flap debulking, etc) are not relevant for the purposes of determining eligibility vis a vis completing oncologic treatment within 6-week to 12 months of enrollment
5. Cancer-free at the time of accrual

   -patients with known indolent malignancies (e.g., non-melanoma skin cancer, low risk thyroid cancer, untreated prostate cancer, etc) would not exclude a patient from the study
6. No planned significant HNC ablative or reconstructive surgery (defined by a postoperative inpatient stay of at least three days) during the study intervention or follow-up period as determined by the HNC oncologic surgeon at the time of study accrual
7. Willingness to be randomized to either BRIGHT or AC
8. IMAGE-HN score ≥ 22

Exclusion Criteria:

1. Inability to speak or read English
2. Pre-existing, ongoing psychotherapy services for any disorder and the participant is not willing to discontinue the prior therapy for the duration of the proposed trial
3. Severe mental illness that would prevent trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
IMAGE-HN | 9 months
  The IMAGE-HN is a 24-item, validated patient-reported outcome measure (PROM) of HNC-related BID. Items are rated on a 5-point Likert scale from 'Never' (0) to 'Always' (4). The total global score is calculated by summing item responses across 21 items (all items except 3, 4, and 19). Total IMAGE-HN scores on the global domain (21 questions) range from 0-84; higher scores indicate worse HNC-related BID. An IMAGE-HN score of > 22 indicates clinically-significant HNC-related BID and a change in IMAGE-HN score of > 9 points is clinically meaningful.

SECONDARY OUTCOMES:
Shame and Stigma Scale-Head and Neck | 9 months
  The Shame and Stigma Scale is a 20-item, validated, unidimensional PROM that measures four domains (shame with appearance, stigma, regret, and social/speech concerns) in patients with HNC over the prior 7 days. Items are rated on a 5-point Likert scale from 'Never' (0) to 'All the time' (4). The total score is calculated by summing the individual responses (except for 4 questions which are reverse scored). Shame and Stigma Scale scores range from 0-80; higher scores reflect worse HNC-related shame and stigma.
PROMIS SF v1.0- Depression 8a | 9 months
  The PROMIS SF v1.0-Depression 8a is an 8-item validated measure developed by the NIH to assess patient-reported negative mood, views of self, and decreased positive affect and engagement. Responses rate the strength of agreement with statements about depressive symptoms using a scale that ranges from 1-5. The total raw score is calculated by summing the individual responses. The PROMIS SF v1.0-Depression 8a raw score ranges from 8-40; a higher score reflects more severe depressive symptoms. The PROMIS SF v1.0-Depression 8a total raw score is translated into a T-score for each participant according to the PROMIS Scoring manual. The T-score provides a standardized score with a mean of 50 and a standard deviation of 10.
PROMIS SF v1.0-Anxiety 8a. | 9 months
  The PROMIS SF v1.0-Anxiety 8a is an 8-item, validated, developed by the NIH to assess patient-reported fear, worry, and hyperarousal. Responses rate the strength of agreement with statements about anxiety symptoms using a scale that ranges from 1-5. The total raw score is calculated by summing the individual responses. The PROMIS SF v1.0-Anxiety 8a raw score ranges from 8-40; a higher score reflects more severe anxiety symptoms. The PROMIS SF v1.0-Anxiety 8a total raw score is translated into a T-score for each participant according to the PROMIS Scoring manual. The T-score provides a standardized score with a mean of 50 and a standard deviation of 10.
Beck Scale for Suicidal Ideation | 9 months
  The Beck Scale for Suicidal Ideation is a 21-item, validated, unidimensional rating scale that measures the current intensity of patients' specific attitudes, behaviors, and plans to commit suicide on the day of the interview. Each item consists of three options graded according to suicidal intensity on a 3-point scale ranging from 0 to 2. The ratings for the first 19 items are summed to yield a total score, ranging from 0 to 38. Higher scores represent more severe suicidal ideation.
PROMIS Short Form (SF) v2.0-Ability to Participate in Social Activities 8a | 9 months
  PROMIS SF v2.0-Ability to Participate in Social Activities 8a is an 8-item, validated, unidimensional measure of patient-reported perceptions of participation in social activities. Items are scored using a 5-point Likert scale from 'Never' (1) to 'Always' (5). The total raw score is calculated by summing the individual responses. The total raw score ranges from 8-40; a higher score reflects more severe inability to participate in social activities. The total raw score is translated into a T-score for each participant according to the PROMIS Scoring manual. The T-score provides a standardized score with a mean of 50 and a standard deviation of 10.
EORTC QLQ-Head Neck 35 Trouble with Social Eating Subscale | 9 months
  The EORTC QLQ-Head Neck 35 Trouble with Social Eating Subscale is a 4-item, validated measure of trouble with social eating for patients with HNC. The subscale is composed of QLQ-H&N35 items 19-22. Items are scored using a 4-point Likert scale from 'not at all' (0) to 'very much' (3). The total score is calculated by summing the individual responses. Total subscale scores range from 0-12; higher scores reflect more trouble with social eating.
EORTC QLQ-HN35 Trouble with Social Contact Subscale | 9 months
  The EORTC QLQ-HN35 Trouble with Social Contact Subscale is a 5-item, validated measure of trouble with social contact for patients with HNC. The subscale is composed of QLQ-H&N35 items 18, 25-28. Items are scored using a 4-point Likert scale from 'not at all' (0) to 'very much' (3). The total score is calculated by summing the individual responses. Total subscale scores range from 0-15; higher scores reflect more trouble with social contact.
Body Image Coping Strategies Inventory (BICSI) | 9 months
  The BICSI is a 29-item, validated measure of the cognitive and behavioral responses to manage threats to body image. BICSI contains three sub-domains; (1) appearance fixing (altering appearance by covering, camouflaging, or correcting the perceived defect), (2) avoidance (an attempt to escape or avert stressful body-image situations), and (3) positive rational acceptance (acceptance of the challenging event and positive self-care or rational self-talk about one's appearance). Items are scored on a 4-point Likert scale from 'Definitely not like me' (0) to 'Definitely like me' (3). The score for each subscale is calculated by summing the values for the individual questions and thus ranges as follows: Appearance fixing (0-30), Avoidance (0-24), and Positive rational acceptance (0-33). For each subscale, higher scores indicate greater reliance on that type of body image coping strategy.
Automatic Thoughts Questionnaire | 9 months
  The Automatic Thoughts Questionnaire is a 15-item, validated, patient-reported measure of negative automatic thoughts. Items are scored using a 5-point Likert scale (1-5). The total score is calculated by summing the individual responses. Total scores range from 15-75; higher scores reflect more negative automatic thoughts.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Pennsylvania State University, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Research materials will include baseline data and study outcomes from trial participants. Data will be raw or minimally processed.
  Data will be available following final database lock, reporting to clinicaltrials.gov, and presentation and publication of study findings describing key primary and secondary objectives.
  De-identified data available will be available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate technology; and (3) a commitment to destroying or returning the data after analyses are completed. All data sharing will comply with laws, regulations, and policies privacy governing data derived from human subjects.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following final database lock, reporting to clinicaltrials.gov, and presentation and publication of study findings describing key primary and secondary objectives. Data will remain available as long as they are useful for the larger research community.
Access Criteria: email to PI (graboyes@musc.edu)

REFERENCES:
- [Derived] Graboyes EM, Maurer SN, Kistner-Griffin E, Armeson K, Starr E, McLeod T, Balliet WE, Doenges J, Slavin-Spenny O, Vanderlan JR, Day A, Pipkorn P, Puram SV, Tam SH, Ruggiero KJ, Sterba KR. Protocol for a multisite, parallel-group, randomized clinical trial comparing a brief tele-cognitive behavioral therapy intervention (BRIGHT) with attention control for the reduction of body image-related distress among head and neck cancer survivors. Contemp Clin Trials. 2025 Jun;153:107888. doi: 10.1016/j.cct.2025.107888. Epub 2025 Mar 24. PMID 40139457

DOCUMENTS (2):
  • Study Protocol (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT05442957/Prot_000.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT05442957/ICF_001.pdf